CLINICAL TRIAL: NCT03780504
Title: A Non-interventional Prospective Observational Study Assessing APRemilast in psOriatic Arthritis in Real-life Clinical Practice in Greek Healthcare Environment. The "APROACH" Study
Brief Title: Apremilast in Psoriatic Arthritis in Real-life Clinical Practice in Greece
Acronym: APROACH
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Genesis Pharma S.A. (Industry)
Collaborators: Celgene (Industry); Amgen (Industry)
Responsible Party: Sponsor
Other Study IDs: GEN-NIS-APR-002
Record Dates: First submitted 2018-12-17; First posted 2018-12-19 (Actual); Last update posted 2021-12-21 (Actual); Status verified 2021-12

CONDITIONS: Psoriatic Arthritis
MeSH Terms: conditions — Arthritis, Psoriatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Following the evidence from the controlled clinical trial setting on the significant clinical benefits of apremilast in the treatment of active PsA, there is a scarcity of real-life evidence on the effectiveness and the beneficial role of apremilast in PsA in routine clinical practice. The present study primarily aims to generate real-world evidence on the impact of apremilast treatment on a broad population of biologic-naïve PsA patients in terms of its clinical effectiveness across the wide spectrum of disease manifestations, as well as its impact on disease burden and HRQoL, in the routine primary care settings of Greece.

DETAILED DESCRIPTION:
Despite tremendous progress achieved in psoriatic arthritis (PsA) over the past 15 years, its management remains challenging due to the clinical heterogeneity and multifaceted nature of the disease. Currently available recommended algorithms for PsA treatment guide clinicians through treatment choices, beginning with conventional synthetic DMARDs after failure of non-steroidal anti-inflammatory drugs (NSAIDs) and local therapy for active disease, followed, if necessary, by a biological DMARD or a targeted synthetic (ts) DMARD. The latter novel category of DMARDs represents recent advances in the treatment options of PsA that aim to overcome the limitations of biological agents that stem by the fact that they have to be administered intravenously or subcutaneously, are very cost intensive for both the patients and the health system, while among them, the immunosuppressive biological agents are also associated with increased risks for infections and certain malignancies. The first approved tsDMARD for the treatment of PsA is apremilast which with an alternative mechanism of action, oral route of administration and favorable safety profile, presents a novel treatment option for PsA that may be appropriate for use early in the treatment algorithm.

Although there is evidence from the controlled clinical trial setting on the significant clinical benefits of apremilast in the treatment of active PsA, and despite the increasing recognition of the value of real-world data as a complementary source to randomized clinical trials, there is a scarcity of real-life evidence on the effectiveness and the beneficial role of apremilast in PsA in routine clinical practice which is partially attributed to the relatively recent advent of apremilast in the market.

In light of the above, the present study primarily aims to generate real-world evidence on the impact of apremilast treatment on a broad population of biologic-naïve PsA patients in terms of its clinical effectiveness across the wide spectrum of disease manifestations, as well as its impact on disease burden and HRQoL, in the routine primary care settings of Greece. This information alongside with collected evidence regarding drug utilisation and safety profile under real-world conditions will strengthen the current state of knowledge in regards to the optimal use of apremilast in this population.

ELIGIBILITY:
Inclusion Criteria:

Patients eligible for inclusion in this study have to meet all of the following criteria:

* Male or female outpatients ≥18 years of age at the time of apremilast treatment onset;
* Patients diagnosed with active peripheral PsA (as per physician's clinical judgement) who have had an inadequate response (to at least one DMARD and within the first 12 months of treatment) or who have been intolerant to a prior DMARD therapy;
* Patients who have been prescribed treatment with apremilast (Otezla®) for PsA, either as a monotherapy or combination therapy with classical systemic DMARD, prior to signed Informed Consent and for whom, if treatment has started, no more than one week has elapsed from treatment initiation to obtaining the signed Informed Consent;
* Patients for whom the decision to prescribe therapy with apremilast according to the locally approved SmPC has already been taken prior to their enrollment in the study and is clearly separated from the physician's decision to include the patient in the current study;
* Patients with available information on the measures needed for the calculation of cDAPSA score at the start of apremilast treatment (i.e., number of swollen and tender joints based on the 66 swollen joint count and the 68 tender joint count, respectively, and patient global assessments of disease activity and pain);
* Patients must be able to read, understand and complete the study specific questionnaires;
* Patients must provide a written Informed Consent prior to inclusion to the study;
* Patients must be able to understand the study procedures and adhere to the study visit schedule.

Exclusion Criteria:

A patient who meets any of the following criteria will be excluded from participation in this study:

* Patients who have a history of exposure to biologic treatment and/or to tofacitinib in PsA;
* Patients that meet any of the contraindications to the administration of the apremilast as outlined in the latest version of the locally approved SmPC;
* Patients who currently receive treatment with any investigational drug/device/intervention or who have received any investigational product within 30 days or 5 half-lives of the investigational agent (whichever is longer) before the start of therapy with apremilast;
* Patients who are currently pregnant, breastfeeding, or planning a pregnancy during the study observation period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population is adult biologic-naïve PsA patients, diagnosed with active peripheral PsA (as per physician's clinical judgement) who have had an inadequate response (to at least one DMARD and within the first 12 months of treatment) or who have been intolerant to a prior DMARD therapy, and who have prescribed treatment with apremilast according to the routine primary care settings of Greece.
Sampling Method: Non-Probability Sample
Enrollment: 170 (Actual)
Dates: Start 2019-04-15 (Actual); Primary Completion 2021-07-20 (Actual); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
evaluate the apremilast impact on peripheral PsA disease activity | at 24 weeks post-treatment onset
  Percentage of patients with active PsA treated with apremilast who will achieve at least 50% improvement in cDAPSA (clinical Disease Activity in Psoriatic Arthritis) baseline score at 24 weeks post-treatment onset

SECONDARY OUTCOMES:
estimate the moderate cDAPSA response rate | at 24 and 52 weeks post-treatment onset
  Percentage of patients with active PsA treated with apremilast who will achieve at least 75% improvement in cDAPSA (clinical Disease Activity in Psoriatic Arthritis) baseline score at 24 weeks and at 52 weeks post-treatment onset, respectively
estimate the major cDAPSA response rate | at 24 and 52 weeks post-treatment onset
  Percentage of patients with active PsA treated with apremilast who will achieve at least 85% improvement in cDAPSA ( (clinical Disease Activity in Psoriatic Arthritis) baseline score at 24 weeks and at 52 weeks post-treatment onset, respectively
classify the study population into the PsA disease activity states | at 52 weeks post-treatment onset
  Percentage of patients in remission (REM), low disease activity (LDA), moderate disease activity (MDA) and high disease activity (HDA) at 52 weeks post-treatment onset, as assessed by DAPSA (Disease Activity in Psoriatic Arthritis) scores, using the cut-off values of ≤4 for REM, >4 and ≤14 for LDA, >14 and ≤28 for MDA and >28 for HDA
evaluate the effect of apremilast treatment on enthesitis (complete resolution) | at 16, 24 and 52 weeks post-treatment onset
  Percentage of patients with enthesitis at baseline who will achieve complete resolution of enthesitis (LEI=0), as assessed by LEI (Leeds Enthesitis Index) score (0-6).
evaluate the effect of apremilast treatment on enthesitis (change in LEI score) | at 16, 24 and 52 weeks post-treatment onset
  Change from baseline in LEI score among the study subpopulation with baseline LEI greater than zero
evaluate the effect of apremilast treatment on dactylitis (complete resolution) | at 16, 24 and 52 weeks post-treatment onset
  Percentage of patients with dactylitis at baseline who will achieve complete resolution of dactylitis (DSS=0), as assessed by the dactylitis severity score (DSS 0-60 for all digits).
evaluate the effect of apremilast treatment on dactylitis (change from baseline) | at 16, 24 and 52 weeks post-treatment onset
  Change from baseline in DSS among the study subpopulation with baseline DSS greater than zero.
evaluate the effect of apremilast treatment on dactylitis (change in digits) | at 16, 24 and 52 weeks post-treatment onset
  Change from baseline in total number of digits affected by dactylitis among the study subpopulation with dactylitis at baseline.
evaluate the effect of apremilast treatment on patients' physical function using the HAQ-DI (change from baseline) | at 16, 24 and 52 weeks post-treatment onset
  Change from baseline in HAQ-DI (Health Assessment Questionnaire-Disability Index) score among the overall study population.
evaluate the effect of apremilast treatment on patients' physical function using the HAQ-DI (percentage of patients) | at 16, 24 and 52 weeks post-treatment onset
  Percentage of patients with HAQ-DI response among the overall study population )(HAQ-DI score: 0-3)

CONTACTS AND LOCATIONS:
Overall Officials: Nikos Antonakopoulos, MD, Study Director — Genesis Pharma S.A.
Locations (1):
- Euromedica Private Clinic, Thessaloniki, Greece

IPD SHARING:
Plan to Share IPD: No